CLINICAL TRIAL: NCT01104298
Title: Randomized, Open, Multicenter, Prospective, Phase II Clinical Trial of Doxorubicin vs. Trabectedin Plus Doxorubicin in the First Line Treatment of Patients With Advanced Non Operable and/or Metastatic Soft Tissue Sarcomas
Brief Title: Doxorubicin vs. Trabectedin Plus Doxorubicin in Non Operable and/or Metastatic STS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis did not show good results for main objective
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-20; 2008-008922-55 (EudraCT Number)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma
Keywords: metastatic STS; Trabectedin; doxorrubicin; soft tissue sarcoma; non operable sarcoma
MeSH Terms: conditions — Sarcoma; Ichthyosis, X-Linked | interventions — Doxorubicin; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Classic Doxorubicin (Adriamycin - Doxorubicin hydrochloride) Presentation: Solution with 10, 20, or 50 mg Doxorubicin Hydrochloride. Excipients: hydrochloric acid and sodium chloride 0.9%, q.s. 25 ml.
  Pharmaceutical form: concentrate for solution for infusion. Route of administration: Intravenous
  Interventions: Drug: Doxorubicin
- Arm B (Experimental): Trabectedin Presentation: vials with trabectedin 1 mg and sucrose 400 mg. Pharmaceutical form: A white or whitish lyophilized powder as concentrate for solution for injection.
  Route of administration: for intravenous use after reconstitution and further dilution.
  Classic Doxorubicin (Adriamycin - Doxorubicin hydrochloride) Presentation: Solution with 10, 20, or 50 mg Doxorubicin Hydrochloride. Excipients: hydrochloric acid and sodium chloride 0.9%, q.s. 25 ml.
  Pharmaceutical form: concentrate for solution for infusion. Route of administration: Intravenous
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Doxorubicin — A maximum of 6 cycles every 3 weeks of doxorubicin monotherapy 75 mg/square meter will be given in the absence of progression or not acceptable toxicity.
  Other Names: Adriamycin
  Arms: Arm A
Drug: Trabectedin — A maximum of 6 cycles every 3 weeks of the combination (Trabectedin 1,1 mg/square meter + doxorubicin 60 mg/square meter) will be given in the absence of progression or not acceptable toxicity.
  Other Names: Yondelis
  Arms: Arm B

SUMMARY:
The proposed investigation intends to explore if the combination of trabectedin and doxorubicin in the first line of treatment of advanced sarcomas obtains better results than doxorubicin monotherapy

DETAILED DESCRIPTION:
The proposed investigation intends to explore if the combination of trabectedin and doxorubicin in the first line of treatment of advanced sarcomas obtains better results than doxorubicin monotherapy.

This proposal arises from the need to bring to the first line of treatment of advanced STS agents that have shown activity in second line. The goal is to improve available standard treatments. Tumors in patients not previously exposed to chemotherapy have not been selected in their biological behavior and they are the best scenario to test antitumor activity of a new anticancer drug.

The combination of drugs with different mechanisms of action may be a clear advantage to obtain better results and potential synergy. On the other hand, the toxicity profiles of both study drugs are different and worsening or summative of adverse effects is not expected.

The purpose of this study is to determine the efficacy of the combination of trabectedin and doxorubicin in comparison with doxorubicin alone in patients with advanced non operable and/or metastatic Soft Tissue Sarcomas (STS).

ELIGIBILITY:
Inclusion Criteria:

* The patient must sign voluntarily the informed consent from before any study test is conducted that is not part of routine patient care, with the knowledge that he/she can abandon the study at any time without this affecting his/her previous care.
* Aged between 18 and 70.
* Pathological diagnosis of non operable and/or metastatic soft tissue sarcoma.
* The following histological subtypes can be included:

  * Undifferentiated pleomorphic sarcoma (previously,malignant fibrous istiocytoma)
  * Leiomyosarcoma
  * Angiosarcoma
  * Liposarcoma
  * Synovial sarcoma
  * Fibrosarcoma
  * Hemangiopericytoma
  * Neurofibrosarcoma
  * Mixofibrosarcoma
  * Unclassified sarcoma
* Measurable disease, according to RECIST criteria
* Performance status 0-2 Eastern Cooperative Oncology Group(ECOG).
* Adequate bone marrow function (hemoglobin > 10 g/dL, leukocytes ≥ 3.000/mm3, neutrophils ≥1.500/mm3, platelets ≥ 100.000/mm3). Patients with plasma creatinine ≤ 1,6 mg/dL, transaminases ≤2.5 times the upper limit of normal (ULN), total bilirubin ≤ upper limit of normal (ULN), CPK ≤ 2.5 times upper limit of normal (ULN), alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN) are acceptable. If the increase of alkaline phosphatase is > 2.5 times the upper limit of normal (ULN), then the alkaline phosphatase liver fraction and/or 5' nucleotidase and/or GGT must be ≤ upper limit of normal (ULN).
* Men or women of child bearing potential should be using an effective method of contraception before entry into the study and throughout the same and for 6 months after ending the study. Women of childbearing potential must have a negative urine pregnancy test before study entry.
* Normal cardiac function with a Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram or Multiple Uptake Gated Acquisition Scan (MUGA).

Exclusion Criteria:

* Previous chemotherapy treatment.
* Previous radiotherapy involving the only localization(s) of measurable tumoral disease.
* Performance status> 2 Eastern Cooperative Oncology Group(ECOG).
* Central Nervous System (CNS) metastases.
* Plasma bilirubin > upper limit of normal(ULN).
* Creatinine > 1.6 mg/dL.
* History of other neoplastic disease with the exception of basalioma or in situ cervical cancer adequately treated.
* Significant cardiovascular disease (for example, dyspnea > 2 NYHA)
* Significant systemic diseases grade 3 or higher on the NCI-CTC version 3.0 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity.
* Uncontrolled bacterial, mycotic or viral infections.
* Women who are pregnant or breast-feeding
* Psychological, familial, social or geographic circumstances that limit the patient's ability to comply with the protocol or informed consent.
* Patients participating in another clinical trial or receiving any other investigational product.
* Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.
* The following histologic subtypes are excluded:

  * Rhabdomyosarcoma
  * Ewing's family of tumors
  * Desmoplastic small round cell tumor
  * Clear cell sarcoma
  * Alveolar sarcoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of the combination of trabectedin and doxorubicin in comparison with doxorubicin alone in patients with advanced non operable and/or metastatic Soft Tissue Sarcomas (STS) | 2012
  To determine the efficacy of the combination of trabectedin and doxorubicin in comparison with doxorubicin alone in patients with advanced non operable and/or metastatic Soft Tissue Sarcomas (STS). To this end, progression free survival will be compared between both groups of treatment.

SECONDARY OUTCOMES:
To determine activity by means of RECIST objective responses in both study arms, trabectedin/doxorubicin combination and the control arm. | 2012
  To determine activity by means of RECIST objective responses in both study arms, trabectedin/doxorubicin combination and the control arm.
To determine the tumor control (response rates plus stabilizations) in both arms of treatment. | 2012
  To determine the tumor control (response rates plus stabilizations) in both arms of treatment.
Overall survival. | 2012
  Overall survival.
To determine activity by tissue changes applying the Choi criteria to Soft Tissue Sarcomas (STS)(see radiological review sub study). | 2012
  To determine activity by tissue changes applying the Choi criteria to Soft Tissue Sarcomas (STS)(see radiological review sub study).
To determine toxicity of trabectedin/doxorubicin combination and the control arm. | 2012
  To determine toxicity of trabectedin/doxorubicin combination and the control arm.
To determine protein and mRNA expression of genes possibly involved in a potential profile of more favorable response or resistance to study drugs and to analyze the prognostic impact of them on predefined efficacy parameters. | 2012
  To determine protein and mRNA expression of genes possibly involved in a potential profile of more favorable response or resistance to study drugs and to analyze the prognostic impact of them on predefined efficacy parameters.
To evaluate genomic instability, as well as protein expression that could influence response/resistance to the study drugs and make a correlation with efficacy endpoints. | 2012
  To evaluate genomic instability, as well as protein expression that could influence response/resistance to the study drugs and make a correlation with efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martin Broto, PhM, Principal Investigator — GEIS; Andres Poveda, Ph.M., Principal Investigator — GEIS
Locations (20):
- Spain (20):
  - Ico Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - ICO Badalona, Badalona
  - H. Clinic Barcelona, Barcelona
  - H. Sant Pau, Barcelona
  - H. Provincial Castellón, Castellon
  - ICO Girona, Girona
  - H. Xeral Cies, Lugo
  - Clinica Puerta Hierro, Madrid
  - H. Clínico. San Carlos, Madrid
  - H. U. La Paz, Madrid
  - H.U. Gregorio Marañon, Madrid
  - H.U. Ramon Y Cajal, Madrid
  - H.U. Clinico de Malaga, Málaga
  - H. de Navarra, Navarra
  - H. C. Asturias, Oviedo
  - H. Son Dureta, Palma de Mallorca
  - H. Univ. Canarias, Santa Cruz de Tenerife
  - H.U. Virgen Del Rocio, Seville
  - Instituto Valenciano de Oncología, Valencia
  - H. Miguel Servet, Zaragoza